CLINICAL TRIAL: NCT03714256
Title: Human Factor Validation of Pediatric Mobility Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Permobil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Per2018P04
Record Dates: First submitted 2018-10-11; First posted 2018-10-22 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Disability Physical
Keywords: Pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Children 6-17 months (Experimental): Device, patient mobility, powered:
  Usability of the pediatric mobility device by both parent/guardian and occupational/physiological therapist, performed according to instructions for use at a one time occasion.
  Interventions: Device: Device, patient mobility, powered
- Children 18 - 36 months (Experimental): Device, patient mobility, powered:
  Usability of the pediatric mobility device by both parent/guardian and occupational/physiological therapist, performed according to instructions for use at a one time occasion.
  Interventions: Device: Device, patient mobility, powered

INTERVENTIONS:
Device: Device, patient mobility, powered — Pediatric mobility device

SUMMARY:
The purpose of this study is to validate the user interface of a pediatric power mobility device by establishing that the product is safe and effective use for the intended users.

DETAILED DESCRIPTION:
The purpose of this study is to validate the user interface of a pediatric power mobility device by establishing that the product is safe and effective use for the intended users. The human factors validation study will be conducted in children with mobility impairments as categorised by Hays (1987) in the age range of 6 months to 36 months under realistic use conditions.The study is an open label, un-blinded, non-randomized study which consists of one visit.

ELIGIBILITY:
Inclusion Criteria:

Primary users:

* Informed consent signed by parents or guardian
* Aged 6-36 months
* Unable to mobilize independently for exploratory play and peer interaction, as categorized by Hays (1987)
* Adequate trunk and head control to remain upright in the device, including regain head control
* Adequate hand/ arm (distal) control to reach for objects in front of them

Secondary users:

* Signed informed consent
* Physiotherapist/Occupational Therapist or parent/guardian of the child included in the test

Exclusion Criteria:

* Primary users:

  * Weight >16 kg/35 Ibs
  * Length >100 cm/39 In
  * Children that lack head control in such a severe manner that they cannot regain control if it is lost
  * Children who do not show awareness of or respond to toys, objects, sounds and/or people in their environment
  * Any other reason, if in the opinion of the investigator, the individual user is not appropriate, or suitable for participation in the test.

Secondary users:

* Hearing/vision loss or limited cognitive skills impacting the ability to take instructions and perform the tasks of the test
* Ability to understand oral and written English as product labelling will in this Human Factor validation test only be available in English
* Any other reason, if in the opinion of the investigator, the individual user is not appropriate, or suitable for participation in the test

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Leire, Study Director — Permobil Group
Locations (3):
- United States (3):
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Oregon State University, Corvallis, Oregon
  - Belmont University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Children 6-17 Months; Children 18 - 36 Months: Device, patient mobility, powered:
  Usability of the pediatric mobility device by both parent/guardian and occupational/physiological therapist, performed according to instructions for use at a one time occasion.
  Device, patient mobility, powered: Pediatric mobility device
Period: Overall Study
Arm/Group | Children 6-17 Months | Children 18 - 36 Months
Started | 14 | 19
Completed | 14 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children 6-17 Months | Children 18 - 36 Months | Total
Number analyzed (Participants) | 14 | 19 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 19 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Use Errors Associated With the Usage of the Device According to Labelling
Description: The tasks in this Human factors validation test, that will be performed by the users are: charge battery and disconnect it, adjust seat and table height, adjust the speed, place the child in device, adjust cushion and other support. The summary of identified errors, captured through observation and interview, will be counted and define the primary outcome
Time Frame: One day
Measure: Number; unit: Errors
Arm/Group | Children 6-17 Months | Children 18 - 36 Months
Number analyzed (Participants) | 14 | 19
Errors | 4 | 2

ADVERSE EVENTS:
Time Frame: During study participation (1 day)
Arm/Group | Children 6-17 Months | Children 18 - 36 Months
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/19
Other Adverse Events (participants affected / at risk) | 0/14 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03714256/Prot_000.pdf